CLINICAL TRIAL: NCT00736281
Title: Sublingual Immunotherapy for Food Allergy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recently published research, this is no longer a novel study.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Robert P. Zitsch III, Department Chair, University of Missouri-Columbia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MU-ENT-1118937
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Food Allergies
Keywords: Sublingual Immunotherapy for Food Allergy; Food Drops for Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Peptides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Food Drops (No Intervention): The patients enrolled in our study will present with food allergy symptoms and diagnostic tests will provide the specific information regarding their food allergies. Once the diagnosis has been made and consent for treatment has been obtained, participants will be randomly assigned to either the group that receives the food allergy intervention with SLIT ( food allergens mixed with 50% glycerin in a vial) or the group that receives the control SLIT (glycerin only). The patients are truly blinded to their treatment because all the SLIT food allergy vials are identical and contain no distinguishing features that could reveal their contents. There is also no difference in taste between a vial containing glycerin and food allergens and a vial containing only glycerin.
- Food Drops (Active Comparator): Group 2 (intervention group) will receive sublingual immunotherapy (escalation followed by maintenance) with vials containing glycerin and the previously diagnosed food allergens (peptides).
  Interventions: Other: Food Drops: Food Allergens (peptides)

INTERVENTIONS:
Other: Food Drops: Food Allergens (peptides) — The patients enrolled in our study will present with food allergy symptoms and diagnostic tests will provide the specific information regarding their food allergies. Once the diagnosis has been made and consent for treatment has been obtained, participants will be randomly assigned to either the group that receives the food allergy intervention with SLIT ( food allergens mixed with 50% glycerin in a vial) or the group that receives the control SLIT (glycerin only). The patients are truly blinded to their treatment because all the SLIT food allergy vials are identical and contain no distinguishing features that could reveal their contents. There is also no difference in taste between a vial containing glycerin and food allergens and a vial containing only glycerin.
  Arms: Food Drops

SUMMARY:
The questions proposed by this study are those of safety and efficacy.

1. Concerning safety: "Are sublingual food drops (SLIT) safe enough to be used for stimulation of natural immune suppression in patients with food allergies?"
2. Concerning efficacy: "Do the drops suppress food allergy enough for patients to eat previously allergic foods with little or no allergic reaction?"

The aim of this trial is to provide systematic collection of data proving the safety and efficacy of food drops in the correction of food allergy. A patient's range of symptoms, which can include but are not limited to fatigue, nausea, vomiting, diarrhea, abdominal pain, and insomnia can be diagnostic indicators of food allergies.

An approach to answering the above questions can be done by a randomized, controlled, blinded study. The design of our study could be reasonable and powerful because this layout limits bias and accounts for placebo effects:

The patients enrolled in our study will present with food allergy symptoms and diagnostic tests will provide the specific information regarding their food allergies. Once the diagnosis has been made and consent for treatment has been obtained, participants will be randomly assigned to either the group that receives the food allergy intervention with SLIT ( food allergens mixed with 50% glycerin in a vial) or the group that receives the control SLIT (glycerin only). The patients are truly blinded to their treatment because all the SLIT food allergy vials are identical and contain no distinguishing features that could reveal their contents. There is also no difference in taste between a vial containing glycerin and food allergens and a vial containing only glycerin. Therefore, a food allergy SLIT randomized-controlled study can be reasonably achieved.

DETAILED DESCRIPTION:
Design:

Randomized-controlled blinded trial to evaluate the safety and efficacy of sublingual immunotherapy for food allergy sufferers. The study will report any adverse events caused by the administration of food allergy drops. Food allergy can manifest itself in many forms including general fatigue, abdominal pain, GERD, nausea, and other symptoms.

End Points:

Comparison between groups 1 and 2 about patient-reported adverse, as well as beneficial, events while on food allergy immunotherapy at 3, 6, 9, 12 months after maintenance dose is achieved (SLIT questionnaire). These comparisons relate to both safety and efficacy issues.

Methodology:

Trial subjects will be identified by their presenting complaints due to ingestion of certain symptomatic foods. Clinical assessment of potential food allergy participants for SLIT will occur according to usual testing standards. All participants will have diagnostic tests (usually RAST analysis and or food challenge techniques) to confirm specific food allergies. Subjects who meet the inclusion criteria will be asked to participate in the study through informed consent. Once consent has been obtained, the subject will be randomly assigned to either the control or the intervention group.

Group 1 (control group) will receive sublingual immunotherapy (escalation followed by maintenance) with vials containing glycerin.

Group 2 (intervention group) will receive sublingual immunotherapy (escalation followed by maintenance) with vials containing glycerin and the previously diagnosed food allergens.

After the offending foods are diagnosed, the subject will be instructed to avoid these foods until they have been on the 9-week escalation doses and the maintenance immunotherapy dose for six months. After this eight-month combined period of escalation and maintenance, the participants will be allowed to reintroduce the known offending foods. In addition, participants will be asked to respond to questionnaires at pre-defined intervals in regards to any adverse symptoms they may have experienced while on maintenance SLIT. These questionnaires will allow us to determine if food drops contribute to adverse events, as well as how effective the drops are at suppressing immune response to previously allergic foods.

Procedures:

At the initial clinic visit, potential subjects will be asked to elaborate on specific food allergy symptoms in order to obtain a better understanding of the food allergies involved. Also, diagnostic tests will be performed based on signs and symptoms and these can include:

1. Clinical History
2. Radioallergosorbent Test (RAST)
3. Oral Food Challenge Participants in the intervention group will receive SLIT with glycerin and individualized food allergens. Subjects in the control group will receive SLIT with glycerin only.

The expected length for an individual's participation is sixteen to eighteen months. This period includes the time between the initial clinic visit and diagnostic work-up, the achievement of SLIT maintenance dose, and the 3,6,9,12 month post-maintenance dose safety questionnaires.

Stopping rules apply to the intervention and placebo groups in the case of an adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic, reproducible symptoms following meals.
2. Multiple food allergies where dietary avoidance is nearly impossible.
3. Patients age 4 and older.
4. Testing to verify food allergies is positive.

Exclusion Criteria:

1. History of anaphylaxis, angioedema, asthma, or life-endangering reactions to certain food products.
2. Children under the age of 4.
3. Previous attempts to treat food allergy (subcutaneous injections).
4. General medical condition that precludes elective therapy (including pregnancy).
5. Inability to follow food allergy SLIT regimen.
6. Autoimmune Disease.
7. Chronic use of steroids.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Validated Questionnaires will be administered to trial participants at 3, 6, 9, 12 months after achieving the maintenance dose of food drops. | safety and efficacy questionnaires administered at 3, 6, 9, 12 months after achieving the maintenance dose of food drops

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schneider, M.S., Study Chair — University of Missouri - Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- University Hospital: Department of Otolaryngology - Head and Neck Surgery, Columbia, Missouri, United States